CLINICAL TRIAL: NCT03861364
Title: Haemodynamic Stability During Induction of General Anesthesia With Propofol and Remifentanil: A Randomized, Controlled, Double-blind Study Comparing Low vs High Propofol Doses.
Brief Title: Hemodynamics During Induction of General Anesthesia With High and Low Propofol Dose.
Acronym: PH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helse Fonna (Other)
Responsible Party: Principal Investigator, Gunnar Helge Sjøen, Overlege, anestesi, Helse Fonna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2019/375; 2019-000958-56 (EudraCT Number)
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Hemodynamics Instability; Anesthesia, General; Anesthesia, Intravenous
Keywords: Cardiac Output (CO); Systolic Blood Pressure (SBP); Systemic Vascular Resistance (SVR); Heart Rate (HR); Stroke Volume (SV); Lithium Dilutional Cardiac Output (LiDCO); Minimal Invasive Hemodynamic Monitor; Propofol; Propolipid
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, double blind.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization made by a person not involved in trial in other ways. Allocation masked in sealed envelopes, stored in a locked cash box only opened by two drug preparing nurses not involved in patient care. Syringe labelled with patient identification (ID) (eg 03Prop). Patient, Care Provider and Investigator blinded for actual concentration of drug. Allocation break after data data wash and processing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Propofol (Active Comparator): High Propofol induction dose
  Interventions: Drug: Propofol
- Low Propofol (Active Comparator): Low Propofol induction dose
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — 2,4 mg/kg
  Other Names: Propolipid
  Arms: High Propofol
Drug: Propofol — 1,4 mg/kg
  Other Names: Propolipid
  Arms: Low Propofol

SUMMARY:
The study objective is to examine if a high propofol dose is non-inferior to a low dose in respect to hemodynamic stability in healthy patients during induction of general anesthesia with propofol and remifentanil.

DETAILED DESCRIPTION:
Typically, one or more adjuvant medications are administered to supplement induction of general anesthesia. When combining anesthetic drugs, the hypnotic effects are often synergistic. Propofol is associated with hypotension and bradycardia and used together with remifentanil or sedative agents it may give synergistic or additive sedative and hemodynamic effects.

Claeys (1988) and Fairfield (1991) examined the cardiovascular effects of propofol 2-2.5 mg/kg induction dose and found significant reductions i SBP and SVR and small changes in CO, SV and HR. De Wit (2016) examined hemodynamic changes in different steady state propofol serum concentrations, and found a dose dependent SBP reduction, reduction in resistance of arterial and systemic circulation and a reduction in mean systemic filling pressures (MSFP) indicative of a reduction in "stressed volumes". The effective dose (ED) 95% for loss of consciousness for propofol was determined to 1.75 mg/kg when used alone, and 1.38 mg/kg when used together with remifentanil 0.25 microg/kg/min (total induction dose 1.75 microg/kg remifentanil) in a study by Koh et al. We want to examine the hemodynamic effects of giving a low (1.4 mg/kg) vs a high (2.4 mg/kg) propofol dose combined with a moderate remifentanil dose (about 1.5 microg/kg).

ELIGIBILITY:
Inclusion Criteria:

* Healthy women
* Age 18-50 years
* Gynecological procedures
* General anesthesia

Exclusion Criteria:

* Pre-existing hypertension
* Diabetes for several years
* Ischemic heart disease
* Cerebrovascular disease
* Heart valve disease
* Verified cardiac arrhythmia
* Anaemia
* Kidney or hepatic disease
* Hypersensitivity for soya, eggs or peanuts
* Pregnancy
* Poor health state
* Illicit substance use
* BMI <20 or >35 kg/m2
* SBP >150 mmHg
* HR >100 beats/min

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure (SBP) | The first 7.5 minutes during induction of general anesthesia
  Relative change of SBP (mmHg)
Heart rate (HR) | The first 7.5 minutes during induction of general anesthesia
  Relative change of HR (beats)

SECONDARY OUTCOMES:
Stroke Volume (SV) | The first 7.5 minutes during induction of general anesthesia
  Relative change of SV (ml/beat)
Cardiac Output (CO) | The first 7.5 minutes during induction of general anesthesia
  Relative change of CO (litre/min)
Systemic Vascular Resistance (SVR) | The first 7.5 minutes during induction of general anesthesia
  Relative change of SVR (dynes-sec/cm5/m2)

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar H Sjøen, MD, Principal Investigator — Helse Fonna
Locations (1):
- Kirurgisk Klinikk-Anestesi, Haugesund, Rogaland, Norway

IPD SHARING:
Plan to Share IPD: Yes
LiDCO-csv raw data and processed data will be made public at the publishers site, and the supporting information by request to the Principal Investigator. Statistical Data Plan is included in Study Protocol.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will be stored for 15 years after end of study, and may be shared during this time frame.
Access Criteria: The data may be shared by contacting the Principal Investigator.

REFERENCES:
- [Background] Koh JC, Park J, Kim NY, You AH, Ko SH, Han DW. Effects of remifentanil with or without midazolam pretreatment on the 95% effective dose of propofol for loss of consciousness during induction: A randomized, clinical trial. Medicine (Baltimore). 2017 Dec;96(49):e9164. doi: 10.1097/MD.0000000000009164. PMID 29245361
- [Background] Claeys MA, Gepts E, Camu F. Haemodynamic changes during anaesthesia induced and maintained with propofol. Br J Anaesth. 1988 Jan;60(1):3-9. doi: 10.1093/bja/60.1.3. PMID 3257393
- [Background] Fairfield JE, Dritsas A, Beale RJ. Haemodynamic effects of propofol: induction with 2.5 mg kg-1. Br J Anaesth. 1991 Nov;67(5):618-20. doi: 10.1093/bja/67.5.618. PMID 1751277
- [Background] de Wit F, van Vliet AL, de Wilde RB, Jansen JR, Vuyk J, Aarts LP, de Jonge E, Veelo DP, Geerts BF. The effect of propofol on haemodynamics: cardiac output, venous return, mean systemic filling pressure, and vascular resistances. Br J Anaesth. 2016 Jun;116(6):784-9. doi: 10.1093/bja/aew126. PMID 27199311
- [Derived] Sjoen GH, Falk RS, Hauge TH, Tonnessen TI, Langesaeter E. Hemodynamic effects of a low versus a high dose of propofol during induction of anesthesia. A randomized trial. Acta Anaesthesiol Scand. 2023 Oct;67(9):1178-1186. doi: 10.1111/aas.14293. Epub 2023 Jun 8. PMID 37291731